CLINICAL TRIAL: NCT01746589
Title: Evaluation Of Visual Outcomes and Contrast Sensitivity After Myopic Wavefront-Optimized Lasik Using the 200 KHZ WAVELIGHT® FS200 Femtosecond Laser and the WAVELIGHT® ALLEGRETTO WAVE® EYE-Q Laser
Brief Title: Visual Outcomes and Contrast Sensitivity After Myopic LASIK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel S. Durrie, MD (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Daniel S. Durrie, MD, President, Durrie Vision
Organization: Durrie Vision (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS200SVR-10-2011
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Myopia
Keywords: LASIK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- myopic LASIK procedure (Other): All subjects will receive bilateral myopic LASIK procedure using the 200 kHz WaveLight® FS200 Femtosecond Laser and the WaveLight® Allegretto Wave® Eye-Q Laser
  Interventions: Device: bilateral myopic LASIK

INTERVENTIONS:
Device: bilateral myopic LASIK — 200 kHz WaveLight® FS200 Femtosecond Laser and the WaveLight® Allegretto Wave® Eye-Q Laser
  Other Names: WaveLight® Femtosecond Laser and WaveLight® Allegretto®

SUMMARY:
Evaluate visual outcomes and contrast sensitivity for subjects undergoing bilateral myopic LASIK procedure using the 200 kHz WaveLight® FS200 Femtosecond Laser and the WaveLight® Allegretto Wave® Eye-Q Laser. The use of advanced technology may decrease the loss of contrast sensitivity and improvement of postoperative visual acuity results.

ELIGIBILITY:
INCLUSION CRITERIA

* Male or female in good general health, 18 years of age or older at the time of the pre-operative examination
* Patient must be able to read, comprehend and willing to give HIPPA and informed consent
* Patient is planning to undergo a bilateral LASIK procedure
* Both eyes must have a manifest refractive error from -1.00 D to -7.00 spherical equivalent with less than or equal to 3.00D of refractive astigmatism as expressed in spectacle minus cylinder form
* Both eyes must have a BSCVA of 20/20 or better
* Both eyes must demonstrate refractive stability confirmed by clinical records, previous glasses, or investigator's discretion.
* Patient must be willing to comply with study dosing and complete the entire course of the study.

EXCLUSION CRITERIA

* A patient with evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye
* A patient seeking monovision
* A patient with a known hypersensitivity to any of the components of the procedural or post-LASIK medications
* A patient requiring the use of any ocular drop(s) and/or medication(s) in either eye during the study period with the exception of ocular drops and/or medications provided by the investigator
* A patient having any surgical procedure within a week preceding the scheduled LASIK surgery
* A patient with any UNCONTROLLED systemic disease (i.e., a potential patient in whom therapy for a systemic disease is not yet stabilized )
* A patient with a history of prior intraocular or corneal surgery (including cataract extraction), active clinically significant ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring) inside the visual axis, or evidence of glaucoma or propensity for narrow angle glaucoma in either eye
* A patient with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results
* A patient with a history of any of the following medical conditions, or any other condition that could affect wound healing: uncontrolled diabetes, collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in Uncorrected Visual Acuity over time postoperatively | Postoperatively immediate (1-3 minutes), 30 minutes, 1 hour, 2 hours, 4 hours, 1 day, and 1 month
  Change in uncorrected visual acuity from baseline, postoperatively, immediately(1-3 minutes) after surgery, 30 minutes, 1 hour, 2 hours, 4 hours, 1 day, and 1 month.

SECONDARY OUTCOMES:
Change in contrast sensitivity postoperatively as compared to baseline | Postoperatively at immediately (1-3 minutes) after surgery, 30 minutes, 1 hour, 2 hours, 4 hours, 1 day and 1 month
  Contrast sensitivity (ability to distinguish between shades of gray) will be measured postoperatively immediately (1-3 minutes) after surgery, 30 minutes,1 hour, 2 hours, 4 hours, 1 day, and 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Durrie Vision, Overland Park, Kansas, United States